CLINICAL TRIAL: NCT07054229
Title: Efficacy and Prognosis of Microwave Ablation Treatment for Papillary Thyroid Microcarcinoma Assessed by Contrast-Enhanced Ultrasound Combined With Genetic and Molecular Diagnostics: A Prospective Observational Study
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Qiyun Ou, Dr., Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2024-512-01
Record Dates: First submitted 2025-06-13; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Microwave Ablation; Contrast-enhanced Ultrasound; Genetic and Molecular Diagnostics; Papillary Thyroid Microcarcinoma
Keywords: microwave ablation; Papillary Thyroid Microcarcinoma; contrast-enhanced ultrasound; Genetic and Molecular Diagnostics
MeSH Terms: conditions — Papillary Thyroid Microcarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- The thyroid nodule was confirmed to be papillary thyroid microcarcinoma by fine-needle aspiration bi: 1. Aged 18-70 years, gender not specified;
  2. Patients with low-risk PTMC receiving initial treatment (meeting all the following criteria: single lesion with a maximum diameter ≤1cm; no cervical lymph node metastasis; no distant metastasis; no extrathyroidal extension; no family history of thyroid cancer; no history of head and neck radiation during childhood);
  3. Patients who have undergone fine-needle aspiration cytology examination of thyroid nodules and 88-gene testing for thyroid cancer before surgery;
  4. Patients voluntarily choose to undergo microwave ablation therapy or surgical resection.
  Interventions: Drug: Contrast enhanced Ultrasound; Genetic: 88-gene panel for thyroid cancer

INTERVENTIONS:
Drug: Contrast enhanced Ultrasound — Contrast Enhanced Ultrasound (CEUS) refers to the observation under ultrasound after the injection of ultrasound contrast agents, such as SonoVue or Lumason.
  Other Names: CEUS
Genetic: 88-gene panel for thyroid cancer — "88-gene panel" refers to a testing combination that includes 88 genes, which are typically associated with the onset, progression, and prognosis of thyroid cancer.

SUMMARY:
In 2016, there were 203,000 new cases of thyroid cancer in China, ranking 7th among all malignant tumours and 4th among women, and showing a rapid growth trend. Papillary thyroid cancer (PTMC) with a diameter of ≤10 mm is the most common type of thyroid cancer, accounting for about 50% to 60% of the total number of cases. Low-risk PTMC is the most common type of thyroid cancer, with low invasiveness and good prognosis. Surgery is the treatment of choice for low-risk PTMC, but it significantly affects the quality of life of patients by affecting the function of the thyroid gland and requiring long-term medication after surgery, as well as having a high incidence of intra- and postoperative complications; there are certain impacts and limitations in the actual treatment. Microwave ablation (MWA) is a therapeutic modality emerging in recent years, which has the characteristics of easy operation, precise positioning, safety and effectiveness, small postoperative damage, fast recovery, fewer complications, and does not affect the aesthetics of the patient, which not only avoids surgical trauma and reduces the anxiety of the patient, but also better preserves the function of the thyroid gland, and its clinical application is becoming more and more widespread. In recent years, the application of microwave ablation in the treatment of PTMC has received more and more attention. Ultrasound, as a first-line examination tool, is accepted by the majority of patients because of its advantages of safety, speed, efficiency, low price and painlessness. Contrast-enhanced ultrasound (CEUS) is a new examination technique developed in recent years, which can provide richer and clearer diagnostic information than conventional ultrasound and colour Doppler ultrasound. Ultrasound contrast agents (e.g. Sonovue, Sonazoid), Sonovue with sulphur hexafluoride microbubbles as the main ingredient and Sonazoid with perfluorobutane microbubbles as the main ingredient, are non-toxic, non-radioactive, do not require allergy testing, and do not have the advantages of liver or kidney toxicity, etc., and are increasingly recognised by the public. Ultrasonography is now widely used in clinical practice as the primary modality for assessing efficacy after thyroid ablation therapy. Molecular diagnosis is one of the most important tools for preoperative diagnosis and invasiveness assessment of thyroid cancer. Common thyroid cancer gene variants include point mutations such as BRAF V600E, RAS, TP53, PIK3CA, and gene integration variants such as CCDC6-RET and ETV6-NTRK3. This project intends to assess the efficacy and prognosis of microwave ablation therapy for micropapillary thyroid cancer by ultrasonography combined with genetic molecular diagnosis, which in turn will assist in clinical treatment decisions.

DETAILED DESCRIPTION:
1.1 Background to the study 1.1.1 Overview of thyroid cancer

Thyroid cancer is the most prevalent malignancy of the endocrine system. Data from the National Cancer Centre show that:

203,000 new cases of thyroid cancer in China in 2016, ranking 7th among all malignant tumours and 4th among women, and showing a rapid growth trend. The most common pathological type of thyroid cancer is papillary thyroid carcinoma (PTC), which accounts for about 85%-90% of the total number of cases, followed by follicular thyroid carcinoma (FTC), medullary thyroid carcinoma (MTC), poorly differentiated thyroid carcinoma (PDTC) and undifferentiated carcinoma (ATC).

1.1.2 Overview of PTMC and its surgical treatment Papillary thyroid carcinoma (PTMC) refers to papillary carcinoma with a diameter of ≤10 mm, whose biological behaviour is relatively mild and disease-specific.

behaviour is relatively mild, and the disease-specific mortality rate is less than 1%. Surgery is currently the treatment of choice for PTMC, and studies have shown that the overall survival rates of PTMC at 10 and 15 years after surgery are 94.6% and 90.7%, respectively.

1.1.3 Clinical treatment of low-risk PTMC Surgery is the preferred treatment option for low-risk PTMC, but there are some disadvantages to surgical treatment, including: surgery affects the thyroid gland, and surgery is not recommended for low-risk PTMC.

These include: surgery affects the function of the thyroid gland and therefore requires long-term medication; there are certain complications during and after surgery; and it affects the quality of life of the patients.

However, surgical treatment also has some disadvantages, including: surgery affects the function of the thyroid gland and requires long-term medication after surgery; there are some complications during and after surgery; and it affects the quality of life of the patients.

Since the 1990s, a clinical study of active surveillance (AS) for low-risk PTMC has been conducted in Japan, and the results showed that it is an optional clinical management modality. However, this clinical management modality has not yet reached a consensus in China due to the uneven distribution of healthcare resources and the fact that patients may not always be in a position to undergo regular review and follow-up, which may lead to consequences such as delayed diagnosis and treatment, and patients' quality of life being affected by anxiety.

With the development of ultrasound and microwave technology, microwave ablation therapy is more and more widely used in papillary thyroid cancer. Studies have shown that microwave ablation therapy has the characteristics of easy operation, precise positioning, high safety, small postoperative damage, fast recovery, few complications and does not affect the aesthetics, which not only avoids the trauma of surgery and reduces the anxiety of patients, but also better preserves the function of the thyroid gland, and its clinical application is becoming more and more widespread.

1.1.4 Ultrasonography Ultrasound, as a first-line examination tool, is accepted by the majority of patients because of its safety, speed, efficiency, low price and painlessness.

It is accepted by the majority of patients. Contrast-enhanced ultrasound (CEUS) is a new examination technique developed in recent years, which can provide richer and clearer diagnostic information than conventional ultrasound and colour Doppler ultrasound. Ultrasound contrast agents (e.g. Sonovue, Sonazoid), Sonovue with sulphur hexafluoride microbubbles as the main ingredient and Sonazoid with perfluorobutane microbubbles as the main ingredient, are non-toxic, non-radioactive, do not require allergy testing, and do not have the advantages of liver or kidney toxicity, etc., and are increasingly recognised by the public. Ultrasonography is now widely used in clinical practice as the primary modality for assessing efficacy after thyroid ablation therapy.

1.1.5 Genetic molecular diagnosis Molecular diagnosis is one of the most important tools for preoperative diagnosis and invasiveness assessment of thyroid cancer. It is now known that the occurrence and development of thyroid cancer are associated with dozens of genetic variants. Common gene variants include BRAF V600E, RAS, TP53, PIK3CA and other point mutations, as well as CCDC6-RET, ETV6-NTRK3 and other gene integration variants.

According to TCGA data published in Nature in 2014, the proportion of PTC patients carrying 'high-risk' mutations such as TERT promoter and TP53 in Western populations is about 10-15%. In the Chinese population, the proportion of patients with 'high-risk' mutations is about 5%-10%, and they are more likely to have cervical lymph node metastasis. These patients may have a higher risk of recurrence or lymph node metastasis after ablative therapy, and ablative therapy is usually not recommended.

The WHO Thyroid Tumour Classification Overview (5th edition), published in 2022, suggests that thyroid cancers less than 1 cm should also be evaluated for aggressiveness in combination with genetic variants, and the Guidelines for the Diagnosis and Management of Thyroid Nodules and Differentiated Thyroid (2nd edition), published in 2023, clearly states that BRAF mutations in combination with mutations in genes such as TERT, PIK3CA, AKT1, and TP53 are indicative of a poor prognosis; any patient carrying BRAF mutations may have a higher risk of recurrence or lymph node metastasis. The Guidelines for the diagnosis and treatment of differentiated thyroid carcinoma (DTC), published in 2021, clearly state that BRAF mutations combined with TERT, PIK3CA, AKT1, TP53 and other mutations indicate a poor prognosis, and that any DTC (differentiated thyroid carcinoma) with a BRAF V600E/RAS mutation combined with TERT or TP53 mutations, or RAS combined with EIF1AX mutations is a 'high-risk' patient for postoperative recurrence.

The European ablation guidelines published in 2021 clearly list high-risk mutations (such as TERT promoter and TP53 mutations) as contraindications to ablation, and there is no relevant recommendation in the field of ablation therapy in China.

1.2 Risk/benefit evaluation This study is an observational, diagnostic study with no obvious potential risks to patients. Evaluating the efficacy and prognosis of microwave ablation therapy for micropapillary thyroid cancer by ultrasonography combined with genetic molecular diagnosis can effectively assist clinical decision-making.

1.2.1 Known potential risks Very few patients may have a potential risk of ultrasound contrast agent allergy.

1.2.2 Known potential benefits Evaluating the efficacy and prognosis of microwave ablation therapy for micropapillary thyroid cancer by ultrasonography combined with genetic molecular diagnosis can assess the risk of recurrent metastasis of the lesion and the presence or absence of recurrent metastasis, and can effectively assist clinical decision-making.

1.2.3 Evaluation of potential risk-benefit This study is a prospective, observational study with low risk and high benefit.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years, gender not specified;
* Patients with low-risk PTMC receiving initial treatment (meeting all the following conditions: single lesion with a maximum diameter ≤1cm; no cervical lymph node metastasis; no distant metastasis; no extrathyroidal extension; no family history of thyroid cancer; no history of head and neck radiation during childhood);
* Patients who have undergone fine-needle aspiration cytology examination of thyroid nodules and 88-gene panel testing for thyroid cancer before surgery;
* Patients voluntarily choose to undergo microwave ablation therapy or surgical resection.

Exclusion Criteria:

* Tumor located in the isthmus of the thyroid;
* Pathological high-risk subtypes (tall cell subtype, columnar cell subtype, diffuse sclerosing subtype, solid/insular subtype, oncocytic subtype);
* Progressive enlargement of the cancer lesion in the short term (increase of more than 3mm within 6 months);
* Pregnant women, lactating women;
* Patients with severe coagulation disorders;
* Patients with contralateral vocal cord dysfunction;
* Patients with contraindications to ultrasound contrast agents;
* Other conditions deemed ineligible for enrollment by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 480 patients who were diagnosed with low-risk papillary thyroid microcarcinoma (PTMC) confirmed by fine-needle aspiration biopsy at Sun Yat-sen Memorial Hospital, Sun Yat-sen University will be included between January 2024 and December 2026.
Sampling Method: Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy and prognosis of microwave ablation therapy for papillary thyroid microcarcinoma | 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, and 60 months postoperatively
  Record the absorption status of the ablated lesion: volume observed by ultrasound imaging after ablation, and assess for the presence or absence of lymph node metastasis.Then, we will compile the postoperative follow-up ultrasound data-including volume measurements and lymph node metastasis status-into an Excel spreadsheet.

CONTACTS AND LOCATIONS:
Overall Officials: Luo, Prof., Study Director — Department of Ultrasound in Medicine, Sun Yat-sen Memorial Hospital, Sun Yat-sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, Analytic Code